CLINICAL TRIAL: NCT02908139
Title: Noninvasive Perioperative Monitoring of Arterial Stiffness, Volume and Nutritional Status in Stable Renal Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Czyżewski, PhD, Medical University of Warsaw
Other Study IDs: PWV/KTx/2016/09
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Arterial Calcification; Aortic Stiffness; High Blood Pressure; Kidney Transplantation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients before kidney transplantation: The study included who had been admitted to the TransplantClinic before kidney transplantation
  Interventions: Device: BR-102 plus PWA; Device: Tanita MC780 MA S

INTERVENTIONS:
Device: BR-102 plus PWA — Monitoring of Arterial Stiffness and Central Aortic Pressure
Device: Tanita MC780 MA S — The device measured the size of total body water (TBW), Extra Cellular Water (ECW), Intra Cellular Water (ICW), fat mass (FM%), visceral fat%, fat free mass (FFM) and basal metabolic rate, (BMR) (kcal).

SUMMARY:
Central blood pressure and pulse wave velocity were measured using a BR 102 Plus PWA device in perioperative time after kidney transplantation

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* no clinical cardiovascular disease during the 6 months preceding entry

Exclusion Criteria:

* not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 40 consecutive patients admitted to Transplant Centre to perform kidney transplantataion were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Differences in pulse wave velocity [m/s] in short postoperative period. | 3 days (one day before kidney transplantation and two days after kidney transplantation)
  Assessment will be performed one day before kidney transplantation and two days after kidney transplantation

SECONDARY OUTCOMES:
Differences in central aortic pressure [mmHg] in short postoperative period. | 3 days (one day before kidney transplantation and two days after kidney transplantation)
  Assessment will be performed one day before kidney transplantation and two days after kidney transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Mazowian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Czyzewski L, Wyzgal J, Czyzewska E, Kurowski A, Sierdzinski J, Truszewski Z, Szarpak L. Assessment of Arterial Stiffness, Volume, and Nutritional Status in Stable Renal Transplant Recipients. Medicine (Baltimore). 2016 Feb;95(6):e2819. doi: 10.1097/MD.0000000000002819. PMID 26871855
- [Result] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Comparative analysis of hypertension and its causes among renal replacement therapy patients. Ann Transplant. 2014 Nov 3;19:556-68. doi: 10.12659/AOT.891248. PMID 25365639
- [Result] Czyzewski L, Wyzgal J, Kolek A. Evaluation of selected risk factors of cardiovascular diseases among patients after kidney transplantation, with particular focus on the role of 24-hour automatic blood pressure measurement in the diagnosis of hypertension: an introductory report. Ann Transplant. 2014 Apr 28;19:188-98. doi: 10.12659/AOT.890189. PMID 24770703